CLINICAL TRIAL: NCT00832884
Title: IV Lacosamide: The Safety of Intravenous Lacosamide
Brief Title: The Safety of Intravenous Lacosamide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Le Bonheur Children's Hospital (Other)
Responsible Party: Principal Investigator, James W. Wheless, Principal Investigator, Le Bonheur Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00570-FB; NCT00720863 (obsolete NCT alias)
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Epilepsy
Keywords: partial; onset; epilepsy; pediatric; lacosamide; partial onset epilepsy; vimpat
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Group 1A (Active Comparator): Lacosamide, IV, 50 mg, once, 30 minutes
  Interventions: Drug: Lacosamide
- Group 2A (Active Comparator): Lacosamide, IV, 100 mg, once, 30 min
  Interventions: Drug: Lacosamide
- Group 3A (Active Comparator): Lacosamide, IV, 150 mg, once, 30 min
  Interventions: Drug: Lacosamide
- Group 4A (Active Comparator): Lacosamide, IV, 200 mg, once, 30 min
  Interventions: Drug: Lacosamide
- Group 1B (Active Comparator): Lacosamide, IV, 50 mg, once, 15 min
  Interventions: Drug: Lacosamide
- Group 2B (Active Comparator): Lacosamide, IV, 100 mg, once, 15 min
  Interventions: Drug: Lacosamide
- Group 3B (Active Comparator): Lacosamide, IV, 150 mg, once, 15 min
  Interventions: Drug: Lacosamide
- Group 4B (Active Comparator): Lacosamide, IV, 200 mg, once, 15 min
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — 0.7 mg/kg (up to maximum of 50 mg) x 5 subjects x 30 minutes; 1.4 mg/kg (up to a maximum of 100 mg) x 5 subjects x 30 minutes; 2.1 mg/kg (up to a maximum of 150 mg) x 5 subjects x 30 minutes; 2.9 mg/kg (up to a maximum of 200 mg) x 5 subjects x 30 minutes.
  0.7 mg/kg (up to a maximum of 50 mg) x 5 subjects x 15 minutes; 1.4 mg/kg (up to a maximum of 100 mg) x 5 subjects x 15 minutes; 2.1 mg/kg (up to a maximum of 150 mg) x 5 subjects x 15 minutes; 2.9 mg/kg (up to a maximum of 200 mg) x 5 subjects x 15 minutes
  Other Names: Vimpat

SUMMARY:
To evaluate the safety of IV Lacosamide in children with partial-onset epilepsy, ages 4-35 years old, inclusive, who are either unable to take oral medication or require intravenous administration of IV Lacosamide.

DETAILED DESCRIPTION:
Lacosamide tablets and intravenous formulations were both approved in the United States in the fall of 2008. Lacosamide is indicated for use as adjunctive therapy in the treatment of partial onset seizure disorder in patients' age seventeen years and older. A parenteral dosage form of Lacosamide is desirable for patients who are temporarily unable to take medication orally. The objective of this study is to evaluate the safety of IV Lacosamide in children with epilepsy, ages 4 to 35 years, who are either unable to take oral medication, or whom parenteral administration of IV Lacosamide is desirable.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of epilepsy and have received anti-epileptic drug therapy prior to initiation of IV Lacosamide
* Patients must have a medical condition in which the parenteral administration of Lacosamide is desirable.
* Patients may be male or female.
* Patients must be 4 years of age or older, and less than age 35 years.
* Patient or his / her legally authorized representative must sign an informed consent form prior to any study specific procedures.

Exclusion Criteria:

* Patients will be excluded from entry into the study if any of the following are true:
* Patient has previously participated in any other intravenous Lacosamide study.
* Patient has status epilepticus within the last 3 months.
* Patient has a history of drug allergy to Lacosamide.
* Patient is pregnant.
* Patient has taken experimental drug within last 30 days.
* Patient with significant hepatic or renal disease.

Ages: 4 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2012-05 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of IV Lacosamide given as a rapid infusion. | one year
  The safety of IV Lacosamide will be assessed in patients in whom parental administration of Lacosamide is warranted.

CONTACTS AND LOCATIONS:
Overall Officials: James W Wheless, MD, Principal Investigator — LeBonheur Children's Medical Center
Locations (1):
- LeBonheur Children's Medical Center, Memphis, Tennessee, United States

REFERENCES:
- [Result] Biton V, Rosenfeld WE, Whitesides J, Fountain NB, Vaiciene N, Rudd GD. Intravenous lacosamide as replacement for oral lacosamide in patients with partial-onset seizures. Epilepsia. 2008 Mar;49(3):418-24. doi: 10.1111/j.1528-1167.2007.01317.x. Epub 2007 Sep 19. PMID 17888078
- [Result] Bialer M, Johannessen SI, Kupferberg HJ, Levy RH, Loiseau P, Perucca E. Progress report on new antiepileptic drugs: a summary of the Fifth Eilat Conference (EILAT V). Epilepsy Res. 2001 Jan;43(1):11-58. doi: 10.1016/s0920-1211(00)00171-6. PMID 11137386
- See also: Study site website — http://www.lebonheur.org